CLINICAL TRIAL: NCT02996136
Title: Assessment of the Clinical Performance of the ARROW-FLU System for the Detection of Influenza A and B in Symptomatic Patients
Brief Title: Assessment of the Clinical Performance of the ARROW-FLU System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sekisui Diagnostics, LLC (Industry)
Collaborators: Beaufort CRO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FLU-001-15
Record Dates: First submitted 2016-12-12; First posted 2016-12-19 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2016-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Swab (Experimental): Nasal Swab
  Interventions: Device: Flu Symptoms
- Nasopharyngeal Swab (Experimental): Nasopharyngeal Swab
  Interventions: Device: Flu Symptoms

INTERVENTIONS:
Device: Flu Symptoms — Flu Symptoms

SUMMARY:
The ARROW-FLU Influenza A&B Test is an in vitro diagnostic immuno-chromatographic assay intended for the qualitative detection of influenza A and influenza B viral nucleoprotein antigens from nasal or nasopharyngeal swab specimens in symptomatic patients. It is intended to aid in the rapid differential diagnosis of influenza A and/or B viral infections. This test is not intended for the detection of influenza C viruses. A negative test is presumptive and it is recommended these results be confirmed by cell culture of an FDA cleared molecular device. Negative results do not preclude influenza virus infection and should not be used as the sole basis for treatment or other management decisions.

DETAILED DESCRIPTION:
This multicenter prospective study will include nasal and nasopharyngeal swabs collected from patients who present with flu-like symptoms and have undergone routine testing for influenza virus strain types A or B. The ARROW-FLU Influenza A&B Test System qualitative results will be compared to a reference method for identification of Influenza A or B to determine the clinical sensitivity and specificity of the device.

The ARROW-FLU Influenza A&B Test system will be performed at CLIA-waived and non-CLIA waived clinical sites. Device operators at CLIA-waived sites will be untrained intended users (e.g. nurses, physician assistants, medical assistants, etc).

A subject's participation in this study will consist of a single visit. Following completion of the informed consent process and a review of Inclusion/Exclusion criteria to determine eligibility, each subject will receive a unique study identification number. After standard of care sampling, two (2) nasal or nasopharyngeal swabs will be obtained from each subject enrolled in the study. The swabs will be collected from the same nostril and alternated in their order of designation for testing (i.e. one for ARROW-FLU Influenza System testing and the other for reference testing. Any swab specimens required for standard of care testing will be collected prior to the specimens for this investigation. Investigational device operators will be blinded to standard of care testing results.

ELIGIBILITY:
Inclusion Criteria:

1. The subject may be of any age and either gender.
2. Preliminary assessment of the subject by the Investigator/Designee should be suggestive of influenza virus infection. Subject should present with an influenza-like febrile respiratory illness defined as both

   * Presentation within that last 48 hours of developing a subjective feeling of being feverish and/or a temperature recorded at the clinic within the last 48 hours of greater than or equal to 100.5 F and
   * At least two of the following symptoms: cough, nasal congestion, rhinorrhea, sore throat, headache, myalgia.
3. Written informed consent must be obtained prior to study enrollment:

   1. A subject who is 18 years or older must be willing to give written informed consent and must agree to comply with study procedures.
   2. The legal authorized representative of a subject who is under the age of 18 must give written informed consent and agree to comply with study procedures. Active written assent should be obtained from children of appropriate intellectual age (as defined by the clinical site's IRB).

Exclusion Criteria:

1. The subject underwent a nasal wash/aspirate as part of standard-of-care (SOC) testing during this study visit.
2. The subject is undergoing treatment currently or within the past seven (7) days of the study visit with either

   * A nasally-administered influenza vaccine (FluMist)
   * Anti-viral medication, which may include but is not limited to Amantadine (Symmetrel), Rimantadine (Flumadine), Zanamivir (Relenza), Oseltamivir (Tamiflu), or Ribavirin.
3. The subject is currently receiving or has received within the past thirty (30) days of the study visit anu experimental biologic, drug, or device including either treatment or therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Performance of the ARROW-FLU Influenza Test | Through study completion, an average of 5 months
  The primary objective of this study is the characterization of the performance of the ARROW-FLU Influenza Test to detect influenza virus strain type A or type B in symptomatic subjects. Qualitative results obtained using the ARROW-FLU Influenza Test will be compared to a reference method or "Gold Standard" (viral culture and/or an FDA cleared molecular assay). Performance data generated will support a 510k submission to FDA for clearance of the assay.

SECONDARY OUTCOMES:
Ability of untrained intended users to effectively perform the ARROW-FLU Influenza Test | Through study completion, an average of 5 months
  The secondary objective of this study is to demonstrate the ability of untrained intended users to effectively perform the ARROW-FLU Influenza A&B Test with insignificant risk of erroneous results. Qualitative results obtained using the ARROW-FLU Influenza Test System will be compared to the reference method for confirmation of results on specimens collected during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Daiva Schmidt, Study Director — Sekisui Diagnostics, LLC
Locations (14):
- United States (14):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Clinical Research of South Florida, Coral Gables, Florida
  - Sunrise Medical Research, Lauderdale Lakes, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Avant Research Associates LLC, Crowley, Louisiana
  - Tristan Medical Research Center / Regeneris Medical, North Attleboro, Massachusetts
  - Children's Mercy, Kansas City, Missouri
  - Accent Clinical Vegas, Las Vegas, Nevada
  - Wake Research Associates, Raleigh, North Carolina
  - Clinical Research Solutions LLC (Ohio), Middleburg Heights, Ohio
  - Clinical Research Solutions LLC (Tennessee), Smyrna, Tennessee
  - Marshfield Clinic, Eau Claire, Wisconsin

IPD SHARING:
Plan to Share IPD: No